CLINICAL TRIAL: NCT06182280
Title: Strategies to Prevent HIV Acquisition Among Transgender Men Who Have Sex With Men (TMSM)
Brief Title: Transmaculine One-on-One and Group Empowerment for Targeted HIV Reduction
Acronym: TOGETHR
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fenway Community Health (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Sari Reisner, ScD, Principal Investigator, Fenway Community Health
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Prevention
Other Study IDs: 1R01MH129175-01A1 (NIH)
Record Dates: First submitted 2023-12-13; First posted 2023-12-26 (Actual); Last update posted 2023-12-26 (Actual); Status verified 2023-12

CONDITIONS: HIV Infections; Adherence, Medication
Keywords: Transgender; Men who have sex with men; pre-exposure prophylaxis; behavioral intervention; HIV prevention
MeSH Terms: conditions — HIV Infections; Medication Adherence; Homosexuality

STUDY DESIGN:
Intervention Model Description: The 2x2 factorial design has two actors: individualized, one-on-one peer navigation (PrEP4T vs none) and group-based behavioral intervention (LS4TM vs none). The comparator is standard-of-care information and resources on HIV prevention and linkage to care.
Who Masked: Investigator, Outcomes Assessor
Masking Description: Blinding will occur at the statistician and investigator levels, but is not possible for participants or staff in the intervention. Participants will be followed for 18 months.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Condition A: Standard of Care (SOC) (No Intervention): SOC will include linkage to the CDC's HIV Prevention Services Locator, a US directory of HIV testing and PrEP services. A Digital Library of HIV prevention, sexual health, and anti-stigma materials (written and video media) will be provided. This content is curated from CDC, Gate Trans Men & HIV Project, UCSF Center for Excellence in Trans Health, and National LGBTQIA+ Health Education Center, among other sources.
- Condition B: Online one-on-one peer navigation (SOC + PrEP4T) (Experimental): PrEP4T is an individualized TMSM-specific intervention consisting of online one-on-one sessions between a peer and a participant. PrEP4T has 9 hours of content: 6 1.5-hour sessions conducted weekly for 6 weeks. Participants will also receive access to the SOC materials.
  Interventions: Behavioral: PrEP4T
- Condition C: Online peer-delivered small group-based behavioral intervention (SOC + LS4TM) (Experimental): LS4TM is a theory-based peer-delivered small group-based behavioral intervention. The LS4TM manualized intervention is comprised of 9 hours of content: 6 2-hour small-group sessions with up to 12 participants per group delivered weekly for 6 weeks. Participants will also receive access to the SOC materials.
  Interventions: Behavioral: LS4TM
- Condition D: Peer-delivered and group-based intervention (SOC + PrEP4T + LS4TM) (Experimental): Both PrEP4T and LS4TM will be delivered to participants. Group D will receive 21 hours of content: 6 2-hour LS4TM sessions and 6 1.5-hour PrEP4T sessions. Group D participants may not receive both interventions simultaneously within 6 weeks.
  Interventions: Behavioral: PrEP4T; Behavioral: LS4TM

INTERVENTIONS:
Behavioral: PrEP4T — PrEP4T is an individualized TMSM-specific intervention adapted from The Fenway Model. PrEP4T consists of online one-on-one sessions between a peer and a participant using a strengths-based case management manualized curriculum. Peer navigators (PNs) share transmasculine community membership with participants and are trained to provide linkages. They use an individualized approach to navigate barriers, apply an assets-based frame to promote resiliencies, and pragmatically leverage these to improve biomedical HIV prevention outcomes. PNs utilize techniques from established behavior change models (e.g., Motivational Interviewing; Transtheoretical Model) in PrEP decision-making.
  Arms: Condition B: Online one-on-one peer navigation (SOC + PrEP4T); Condition D: Peer-delivered and group-based intervention (SOC + PrEP4T + LS4TM)
Behavioral: LS4TM — LS4TM is a theory-based peer-delivered small group-based behavioral intervention to reduce HIV risk and address mental health-related effects of stigma for TMSM. Groups will be led by trained peer navigator staff and comprise no more than 10 participants per cohort.
  Arms: Condition C: Online peer-delivered small group-based behavioral intervention (SOC + LS4TM); Condition D: Peer-delivered and group-based intervention (SOC + PrEP4T + LS4TM)

SUMMARY:
Transgender masculine and gender diverse people who have sex with men (TMSM) have an increased risk of HIV and face unique barriers engaging in prevention services. Digitally delivered support interventions addressing HIV prevention barriers delivered by peers in one-on-one or small-group settings may be effective at increasing PrEP engagement. This study examines the independent and combined effects of individual and group-based peer-support interventions on PrEP outcomes. Participants will be randomly assigned to receive: (i) standard-of-care HIV prevention information, (ii) a one-on-one healthy lifestyle intervention tailored for transgender masculine people, (iii) a peer-group based healthy lifestyle intervention for transgender masculine people, or (iv) both the one-on-one and group-based interventions delivered together. The hypotheses are that the individual group-based interventions will result in higher PrEP uptake and persistence than the standard of care and that the combined interventions will be more effective than receiving one individual intervention.

DETAILED DESCRIPTION:
This study will comprise a digitally delivered, open-label randomized 2x2 factorial trial (1:1:1:1 randomization) of peer-delivered HIV prevention strategies. The 2x2 factorial design has two actors: individualized, one-on-one peer navigation (PrEP4T vs none) (Condition B) and group-based behavioral intervention (LS4TM vs none) (Condition C). The trial will compare the efficacy of the interventions to increase PrEP uptake.

Participants in Conditions B and C will receive 6 weeks of their assigned intervention in addition to SOC. Participants in Condition D will be assigned to receive both interventions which may not occur simultaneously. Follow-up will continue another 15 months after the intervention ends to assess effects. In the final 6 months of this 5 years study, PrEP4T and LS4TM will be offered to all participants, regardless of study group assignment. We will ask which intervention participants prefer and gather implementation data.

Randomization and intervention allocation will be automated and computer-generated through an electronic system; the allocation sequence will be concealed. Stratified randomization by race/ethnicity (BIPOC and white) and Movement Advancement Project state LGBTQ equality policy tally (high, medium, or fair overall policy tally as of October 2023, and low or negative overall policy tally as of October 2023) will ensure balance across groups and allow subgroup analyses.49 Blinding will occur at the statistician and investigator levels, 50 but is not possible for participants or staff in the intervention. Participants will be followed for 18 months.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or over
* Assigned female sex at birth
* Identifies as a man, trans man, or another transmasculine identity
* Has had sex with a partner assigned male sex at birth with a flesh penis in the last 3 months
* Has access to a smartphone or computer with internet access
* Is HIV-uninfected
* Resides in one of the Ending the Epidemic targeted geographic hotspots in the United States
* Willing and able to provide informed consent in English
* Meets CDC guidelines for PrEP indications in the last 3 months (adapted for TMSM) including:
* Condomless receptive vaginal/frontal or anal sex with a partner assigned male at birth with a flesh penis
* Sharing needles or syringes for illicit drug use and/or hormones
* Self-reported anogenital sexually transmitted infection diagnosis

Exclusion Criteria:

* Less than age 18
* Not assigned female sex at birth
* Does not identify as a man, trans man, or another transmasculine identity
* Does not have access to a smartphone or computer
* Is living with HIV (HIV positive)
* Does not reside in one of the Ending the Epidemic geographic hotspots in the United States
* Will not or cannot provide written informed consent in English
* Does not meet the trans-adapted CDC guidelines for PrEP indications

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Identify as a man, trans man, or another transmasculine identity
Enrollment: 375 (Estimated)
Dates: Start 2024-01 (Estimated); Primary Completion 2026-07 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
PrEP uptake | 18 months
  Uptake of new PrEP prescriptions during the study intervention and follow-up period as measured by biomarker sampling collected by dried blood spots.

SECONDARY OUTCOMES:
PrEP adherence and persistence | 18 months
  Measurement of PrEP use or disuse across the intervention and follow-up periods as measured by biomarker sampling collected by dried blood spots.

CONTACTS AND LOCATIONS:
Locations (1):
- Fenway Community Health, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Reisner SL, Scheim AI, Cole SW, Wirtz AL, Poteat T, Mimiaga MJ, Marzinke MA, Meyer AI, Smith K, Pletta DR, Mayer KH. Transgender Men and Transmasculine One-on-One and Group-Delivered Empowerment for Targeted HIV Reduction (TOGETHR) Study: Protocol for a Digital Factorial Randomized Controlled Trial. JMIR Res Protoc. 2025 Oct 20;14:e76831. doi: 10.2196/76831. PMID 41115262